CLINICAL TRIAL: NCT04892615
Title: The Safety Research of Timing of the Removal of Abdominal Drains After Pancreatic Surgery ： Results of a Prospective Randomized Clinical Trial
Brief Title: he Safety Research of Timing of the Removal of Abdominal Drains After Pancreatic Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Xian-Jun Yu (Other)
Responsible Party: Sponsor-Investigator, Xian-Jun Yu, President of Pancreatic Cancer Institute, Fudan University
Organization: Fudan University (Other)
Other Study IDs: CSPAC-34
Record Dates: First submitted 2021-05-15; First posted 2021-05-19 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Safety Issues

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort A: The drainage tube was removed on the 5th day after surgery.
  Interventions: Device: drainage tube was removed on 5th days after surgery.
- Cohort B: The drainage tube was removed on the 7th day after surgery.
  Interventions: Device: drainage tube was removed on 7th days after surgery.

INTERVENTIONS:
Device: drainage tube was removed on 5th days after surgery. — drainage tube was removed on 5th days after surgery.
  Groups: Cohort A
Device: drainage tube was removed on 7th days after surgery. — drainage tube was removed on 7th days after surgery.
  Groups: Cohort B

SUMMARY:
Randomized, open, single-center, controlled prospective studies were designed to obtain reliable level I evidence in evidence-based medicine.Based on the premise of at least a 6-fold reduction in pancreatic fistula, as observed by Kawai et al after early drainage.Considering the overall incidence of pancreatic fistula after standard pancreatectomy at our center (approximately 20%), we would expect this complication to occur in approximately 3.4% of cases in Group A.α was set as 0.05 and β was set as 0.2 (efficacy was 80%), indicating that the total number of study subjects was at least 114 patients (at least 57 patients in the experimental group and 57 patients in the control group).

ELIGIBILITY:
Inclusion Criteria:

* ECOG 0-2;
* The amylase value in the drainage tube of patients receiving pancreaticoduodenectomy or distal pancreatectomy was lower than 5000 IU/L on the first day after surgery;
* postoperative drainage tube placement;
* Patients with no obvious contraindication to surgery;
* Expected postoperative survival ≥3 months;

Exclusion Criteria:

* Pancreaticoduodenectomy and pancreaticogastric anastomosis were performed;
* Suspicion or abdominal bleeding within 5 days after surgery;
* suspected biliary and intestinal fistula within 5 days after operation;
* On the fifth day after the operation, abdominal CT reexamination showed local effusion with a depth greater than 3cm.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prepare for elective pancreatic surgery, including laparoscopic or open pancreaticoduodenectomy and distal pancreaticocaudal body resection;
Sampling Method: Probability Sample
Enrollment: 114 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2024-01-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of postoperative pancreatic fistula and abdominal infection; | 3month
Severity of complications (duration of postoperative hospital stay) was assessed by Dindo Clavien classification. | 3month

CONTACTS AND LOCATIONS:
Overall Officials: Xianjun F Yu, Principal Investigator — Fudan University
Locations (1):
- Xianjun Fudan Yu, Shanghai, Sahnghai, China

IPD SHARING:
Plan to Share IPD: Undecided